CLINICAL TRIAL: NCT00767442
Title: Least Invasive Nonlinear Light Microscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Wen-Jeng Lee, NTUH
Other Study IDs: 200806021D
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Oral Leukoplakia; Oral Cancer
MeSH Terms: conditions — Leukoplakia, Oral; Mouth Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Health volunteer
- 2: Patient with suspected oral mucosa lesion

SUMMARY:
Evaluate the ability to image oral mucosa in healthy volunteer by nonlinear microscopy

ELIGIBILITY:
Inclusion Criteria:

* Health volunteer
* Patient with suspected oral mucosa lesion

Exclusion Criteria:

* Active infectious disease
* Inability to cooperate

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Clinics
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jeng Lee, M.D., Principal Investigator — NTUH
Locations (1):
- National Taiwan University Hospital, Taipei, TW, Taiwan